CLINICAL TRIAL: NCT05244616
Title: Validation of the Arabic Version of the Postoperative Quality of Recovery Score 15 (Qor-15Ar)
Status: Completed | Type: Observational
Sponsor: Avicenna Military Hospital (Other)
Responsible Party: Principal Investigator, Younes Aissaoui, MD, Head of surgical intensive care unit, Avicenna Military Hospital
Other Study IDs: QoR-15Ar-AMH
Record Dates: First submitted 2022-02-15; First posted 2022-02-17 (Actual); Last update posted 2022-09-08 (Actual); Status verified 2022-09

CONDITIONS: Postoperative Recovery
Keywords: postoperative recovery - Quality of recovery score 15 - Arabic

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: arabic version of the postoperative Quality of Recovery Score 15 — The Arabic version of the Postoperative Quality of Recovery Score 15 to be completed twice by the patients: once preoperatively and once within 24 to 48 hours postoperatively.

SUMMARY:
Anesthesia practice is not only centered on the patient's safety and well-being through the perioperative period but also on enhancing his overall recovery experience. This study aims to provide an adapted questionnaire for the Arabic-speaking population as a measuring tool of the quality of recovery after surgery.

DETAILED DESCRIPTION:
With the increasing number of anesthesia procedures performed every year, the concept of rapid rehabilitation after surgery has become a primary goal of the perioperative management of patients. This postoperative recovery concerns not only the physical aspect but also encompasses the general concept of well-being and enhancement of the patient's experience. There are many tools to assess postoperative recovery. However, none has been validated within the Moroccan surgical population.

The Qor-15 (Quality of Recovery) score is a scale for measuring postoperative recovery. It was developed in 2013 by Myles et al and has been validated in a widely variable population [1]. It includes 15 items, each rated from 0 to 10. Our objective is to validate the Arabic version of the QOR-15Ar within a Moroccan surgical population.

ELIGIBILITY:
Inclusion Criteria:

* patients admitted for an emergency or elective surgical procedure.

Exclusion Criteria:

* patients under 18 years old
* a weak understanding of the Arabic language
* intracranial Surgery
* underlying psychiatric pathology compromising the completion of the questionnaire
* the presence of life-threatening postoperative complications (e.g. hemorrhagic shock, etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients undergoing elective or emergency surgery admitted at Avicenna Military Hospital
Sampling Method: Non-Probability Sample
Enrollment: 126 (Actual)
Dates: Start 2022-02-16 (Actual); Primary Completion 2022-07-02 (Actual); Study Completion 2022-07-02 (Actual)

PRIMARY OUTCOMES:
Psychometric properties of of the Arabic version of the postoperative quality of recovery score 15 (Qor-15Ar) | Preoperatively and 24 to 48 hours postoperatively.
  The psychometric qualities of the Arabic version of the QoR-15Ar include reliability, validity, and sensitivity to change.
Acceptability and feasibility of the Arabic version of the postoperative quality of recovery score 15 (Qor-15Ar) | Preoperatively and 24 to 48 hours postoperatively.
  The acceptability and feasibility of the questionnaire will be assessed by the participation rate and the time required to complete the questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Avicenna Military Hospital, Marrakesh, Marrakesh Tensift El Haouz, Morocco

IPD SHARING:
Plan to Share IPD: Yes
The data that support the findings of this study will be available from the investigators upon reasonable request.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Immediately following the end of the study .
Access Criteria: Anyone who wish to access the data.